CLINICAL TRIAL: NCT04221165
Title: Opioid Therapy vs Multimodal Analgesia in Head and Neck Cancer: A Randomized Clinical Trial
Brief Title: Opioid Therapy vs Multimodal Analgesia in Head and Neck Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Collaborators: Ontario Institute for Cancer Research (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: OPTIMAL HN
Record Dates: First submitted 2020-01-06; First posted 2020-01-09 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2024-02

CONDITIONS: Head and Neck Cancer; Radiation-Induced Mucositis
Keywords: Pain; Analgesia
MeSH Terms: conditions — Head and Neck Neoplasms; Pain; Agnosia | interventions — Analgesics, Opioid

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Opioid Analgesia (Active Comparator): Opioids will be prescribed as per institutional standards. Examples of opioids are morphine and hydromorphone.
  Interventions: Drug: Opioids
- Multimodal Analgesia (Experimental): Pregabalin (50 mg to 300 mg, oral, twice daily), acetaminophen (1000 mg, oral, 3 times per day), naproxen 250 mg to 500 mg, oral, twice daily), and pantoprazole magnesium (40 mg, oral, daily)
  Interventions: Drug: PAiN - multimodal analgesia

INTERVENTIONS:
Drug: Opioids — Opioids will be prescribed as per institutional standards.
  Arms: Opioid Analgesia
Drug: PAiN - multimodal analgesia — PAiN: Pregabalin, Acetaminophen, Naproxen, pantoprazole magnesium
  Arms: Multimodal Analgesia

SUMMARY:
The purpose of this study is to compare the daily pain level scores for patients taking opioids alone for pain relief, compared with those treated by multimodal analgesia with three medications: pregabalin, naproxen, and acetaminophen, with the ability to switch over to opioid medications if needed. In addition to pain level scores, this study will compare opioid use (length of time and doses taken), quality of life, admissions to hospital, feeding tube requirements, weight loss, and treatment interruptions between these two analgesic regimens.

DETAILED DESCRIPTION:
A significant proportion of patients undergoing radiotherapy alone or chemotherapy and radiotherapy together for their head and neck cancer experience mucositis, which is severe pain in the mouth and throat caused by radiation treatment. Patients often enter a cycle of pain, difficulty swallowing, malnourishment, and reduced quality of life. This may translate into decreased oral intake requiring a feeding tube, and radiation or chemotherapy treatment breaks, which reduce the chance of tumour control and cure.

Currently, opioid therapy is the cornerstone of head and neck cancer pain management. Although effective for pain relief, opioids can have side effects.

As an alternative to opioid treatments, "multimodal analgesia" is a treatment using medications from different classes with different mechanisms of action. Examples of analgesic medications used for multimodal analgesia include medications similar to acetaminophen or ibuprofen, and others.

The primary purpose of this study is to compare pain level scores of patients taking opioids versus patients taking multimodal analgesia.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 or older
* Willing to provide consent
* Histologically confirmed mucosal head and neck malignancy
* Undergoing chemoradiotherapy or radiotherapy alone with a planned total radiation dose of 50 Gray (Gy) or greater
* Eastern Co-operative Oncology Group (ECOG) performance status 0-2
* Life expectancy > 6 months
* Onset of 4/10 pain on the 11-Numeric Rating Scale that is localized to the mucosa of the mouth or throat, before or during radiation treatment, that is not caused by a current oral candidiasis infection.
* Ability to take pills, either by mouth or crushed via NasoGastric (NG) tube or Gastrostomy tube (G-tube)
* Ability to complete the study questionnaires and pain diary
* Ability to sign consent without requirement for a substitute decision maker

Exclusion Criteria:

* Skin and salivary gland malignancies
* High daily opioid use at time of enrollment (defined as 30 mg oral morphine equivalent dose or higher)
* Concurrent second active malignancy
* Pregnant or lactating women
* Psychological disorder requiring pharmacologic treatment
* Regular systemic steroid use
* Regular anticonvulsant or antidepressant use
* Renal Impairment (defined as creatinine clearance < 60 mL/min)
* Liver Dysfunction (defined as total bilirubin > 34.2 µmol/L)
* Documented true allergy to acetaminophen, NSAIDs, pregabalin or opioids
* History of upper gastrointestinal bleed
* Known bleeding disorder
* History of or current substance use disorder

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2020-08-04 (Actual); Primary Completion 2023-09-15 (Actual); Study Completion 2023-09-15 (Actual)

PRIMARY OUTCOMES:
Average Pain Rating measured on the 11 Numeric Rating Scale | Approximately 2 years and 3 months
  Average pain rating during the last 7 days of radiation therapy, as reported by the patient on the 11-Numeric Rating Scale (11-NRS). On the 11-NRS, zero (0) is no pain, and ten (10) is the worst possible pain.

SECONDARY OUTCOMES:
Average Weekly Opioid Use | Approximately 2 years and 4 months
  The average weekly total opioid dose in oral morphine equivalent dosing from randomization to 6 weeks after completion of radiation treatment.
Duration of Opioid Requirement | Approximately 2 years and 6 months
  The time from the start of opioid treatment after randomization to the time of stopping opioid analgesia, in days.
Average Daily 11-Numeric Rating Scale for Pain | Approximately 2 years and 4 months
  Average pain rating from the time of randomization until 6 weeks after completion of radiation treatment, as reported by the patient on the 11-Numeric Rating Scale (11-NRS). On the 11-NRS, zero (0) is no pain, and ten (10) is the worst possible pain.
Quality of Life as measured by the European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire-C30 (EORTC QLQ-C30) | Approximately 24 months, 27 months, and 30 months
  Quality of life, as reported by the patient, will be assessed using the EORTC QLQ-C30 validated questionnaire. Responses regarding function and symptoms are on a scale of 1 (not at all) to 4 (very much). Also included are questions about overall health and quality of life. Responses are on a scale of 1 (very poor) to 7 (excellent).
Quality of Life as measured by the European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire - Head & Neck 43 (EORTC QLQ-HN 43) | Approximately 24 months, 27 months, and 30 months
  Quality of life, as reported by the patient, will be assessed using the EORTC QLQ-HN 43 validated questionnaire. Responses regarding symptoms or problems are on a scale of 1 (not at all) to 4 (very much). This questionnaire is specifically for patients with head and neck cancer.
Average Weekly Opioids Dispensed | Approximately 2 years and 4 months
  The average weekly total opioid dose dispensed by the pharmacy in oral morphine equivalent dosing from randomization to 6 weeks after completion of radiation treatment.
Hospital Admissions | Approximately 27 months and 30 months
  Hospital admissions for febrile neutropenia, serious infection requiring intravenous antibiotics, gastrointestinal bleeding, myocardial infarction, stroke, and acute kidney injury.
Time to Feeding Tube Insertion | Approximately 2 years and 3 months
  The time to feeding tube insertion (e.g. gastrostomy-tube or nasogastric-tube) after randomization, in days.
Weight Loss | Approximately 2 years and 3 months
  Weight loss from randomization to the end of radiation treatment.
Rates of Common Terminology Criteria for Adverse Events Toxicities | Approximately 2 years and 6 months
  Rates of pre-specified Common Terminology Criteria for Adverse Events (CTCAE) toxicities.
Treatment Interruptions | Approximately 2 years and 6 months
  Number of participants with radiation of chemotherapy treatment interruptions.
Death | Approximately 2 years and 6 months
  Number of participants who die during or within 3 months after completion of radiation treatment.

CONTACTS AND LOCATIONS:
Overall Officials: David Palma, MD, Principal Investigator — London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's
Locations (1):
- London Regional Cancer Program of the Lawson Health Research Institute, London, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Elad S, Yarom N. The Search for an Effective Therapy and Pain Relief for Oral Mucositis. JAMA. 2019 Apr 16;321(15):1459-1461. doi: 10.1001/jama.2019.3269. No abstract available. PMID 30990535
- [Background] Lalla RV, Bowen J, Barasch A, Elting L, Epstein J, Keefe DM, McGuire DB, Migliorati C, Nicolatou-Galitis O, Peterson DE, Raber-Durlacher JE, Sonis ST, Elad S; Mucositis Guidelines Leadership Group of the Multinational Association of Supportive Care in Cancer and International Society of Oral Oncology (MASCC/ISOO). MASCC/ISOO clinical practice guidelines for the management of mucositis secondary to cancer therapy. Cancer. 2014 May 15;120(10):1453-61. doi: 10.1002/cncr.28592. Epub 2014 Feb 25. PMID 24615748
- [Background] Mirabile A, Airoldi M, Ripamonti C, Bolner A, Murphy B, Russi E, Numico G, Licitra L, Bossi P. Pain management in head and neck cancer patients undergoing chemo-radiotherapy: Clinical practical recommendations. Crit Rev Oncol Hematol. 2016 Mar;99:100-6. doi: 10.1016/j.critrevonc.2015.11.010. Epub 2015 Dec 3. PMID 26712589
- [Background] Alfieri S, Ripamonti CI, Marceglia S, Orlandi E, Iacovelli NA, Granata R, Cavallo A, Pozzi P, Boffi R, Bergamini C, Imbimbo M, Pala L, Resteghini C, Mirabile A, Locati LD, Licitra L, Bossi P. Temporal course and predictive factors of analgesic opioid requirement for chemoradiation-induced oral mucositis in oropharyngeal cancer. Head Neck. 2016 Apr;38 Suppl 1:E1521-7. doi: 10.1002/hed.24272. Epub 2016 Feb 5. PMID 26849016
- [Derived] Zayed S, Lang P, Read N, Correa RJM, Mutsaers A, Goodman CD, D'Angelo K, Kieraszewicz K, Vanwynsberghe D, Kingsbury-Paul A, Crewdson K, Neeb J, Carreau C, Winquist E, Kuruvilla S, Stewart P, Moulin DE, Warner A, Palma DA. Opioid therapy vs. Multimodal analgesia in head and neck cancer (OPTIMAL-HN): Results of a randomized clinical trial. Radiother Oncol. 2025 May;206:110831. doi: 10.1016/j.radonc.2025.110831. Epub 2025 Mar 5. PMID 40054624
- [Derived] Zayed S, Lang P, Mendez LC, Read N, Sathya J, Venkatesan V, Moulin DE, Warner A, Palma DA. Opioid therapy vs. multimodal analgesia in head and neck Cancer (OPTIMAL-HN): study protocol for a randomized clinical trial. BMC Palliat Care. 2021 Mar 19;20(1):45. doi: 10.1186/s12904-021-00735-0. PMID 33740977